CLINICAL TRIAL: NCT06545279
Title: Success Rate, Child and Parent Acceptance of Modified Hall Crowns Versus Conventional Hall Crowns:A Randomized Clinical Trial
Brief Title: The Success Rate and Acceptability of Conventional and Modified Hall Crowns Among Children and Parents
Acronym: Hallcrowns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20230328
Record Dates: First submitted 2024-06-09; First posted 2024-08-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Paediatric Dentistry; Dental Caries in Children; Dental Treatment
Keywords: Hall crown; Stainless steel crowns; Minimally invasive caries management; biologic caries management; paediatric dentistry

STUDY DESIGN:
Intervention Model Description: Split mouth randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Crown Technique (Experimental): preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal or tooth preparation in one side.
  Interventions: Procedure: Hall Crown Technique
- Modified Hall Technique (Experimental): preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal but with prior interproximal slicing on other side
  Interventions: Procedure: Modified Hall Technique

INTERVENTIONS:
Procedure: Hall Crown Technique — preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal or tooth preparation.
  Arms: Hall Crown Technique
Procedure: Modified Hall Technique — preformed metal crowns (PMCs) cemented with no local anesthesia, caries removal or tooth preparation but with interproximal slicing.
  Arms: Modified Hall Technique

SUMMARY:
This is a clinical trial that aims to compare the success rate, child and parent acceptance of conventional Hall crown technique (CHT) to modified Hall crown technique (MHT)in treating carious primary molars. Eligible children will receive CHT on one side and MHT on the other side. The time interval between both visits will be 1-2 weeks.Patients demographics and pain history will be recorded and pre-operative radiographs will be taken. An observer will assess and record the child's pain perception during each treatment visit. Time taken for each procedure will be recorded by the research assistant each visit prospectively from the moment the child sits on the dental chair till the end of procedure. Parental preference and child acceptance for each procedure will be recorded after treatment is finished using parent and child questionnaire. Clinical follow up will be conducted at 3,6 and 12 months to assess and compare the success rates of both techniques. Radiographs will be taken at 12 months to evaluate and compare radiographic success.

DETAILED DESCRIPTION:
This is a split mouth randomized clinical trial that aims to compare the success rate, child and parent acceptance of conventional Hall crown technique (CHT) to modified Hall crown technique (MHT)in treating carious primary molars. Eligible children will receive CHT on one side and MHT on the other side. The time interval between both visits will be 1-2 weeks.Patients demographics and pain history will be recorded and pre-operative bitewings will be taken. An observer (research assistant who will be trained, calibrated, and blinded to the treatment used) will assess and record the child's pain perception during treatment visit. Time taken for each procedure will be recorded by the research assistant each visit prospectively from the moment the child sits on the dental chair till the end of procedure. Parental preference and child acceptance for each procedure will be recorded after treatment is finished using parent and child questionnaire. Clinical follow up will be conducted at 3,6 and 12 months to assess and compare the success rates of both techniques.Bitewings will be taken at 12 months to assess for crown fit and radiographic pathology.

ELIGIBILITY:
Inclusion Criteria:

* Fit and healthy (ASA 1) children.
* 4-9 years old children.
* Bilateral ICDAS (1, 2, 3 or 4) class I or II carious lesions on primary molars matched for tooth type.
* Teeth with vital pulp with no signs or symptoms of irreversible pulpitis, necrosis, or an abscess.
* No tenderness to percussion, or pathological mobility.
* Prior bitewings must be available showing no radiographic evidence of interradicular radiolucency or caries reaching pulp.
* Contact point is closed.
* Patient has good level of cooperation for the intended procedure.
* Parents consented for their children to be included in the study.

Exclusion Criteria:

* Child with systemic illness (ASA 2,3,4).
* Unmatched carious lesions on primary molars.
* Teeth with deep caries (ICDAS score5 or 6) requiring pulp therapy.
* Irreversible pulpitis or pulp necrosis.
* Pathological mobility.
* Prior bitewings are unavailable.
* Contact point is open.
* Patient has poor level of cooperation for the intended procedure.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | during intervention
  child's pain perception during intervention recorded by research assistant using sound,eyes and motor (SEM) scale
Child discomfort score | immediately following intervention
  Self-reported Child's discomfort after intervention using Wong-Baker FACES Pain Rating Scale
Child acceptance of treatment | immediately following intervention
  Self-reported child acceptance using questionnaire
Parent acceptance of treatment | immediately following intervention
  Parental acceptance using questionnaire
Rate of clinical success | 6,12 months
  Absence of pain symptoms/ dental abscess requiring pulp therapy or extraction ,assessed through taking pain history and clinical examination
Rate of radiographic Success | 12 months
  Absence of radiographic pathology in the root and the bone in the inter-radicular area.

SECONDARY OUTCOMES:
Time taken for intervention | during intervention
  Time taken for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Areej YA Alqadi, Dr, Principal Investigator — Jordan University of Science and Technology; Ola Al-Batayneh, Prof, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No